CLINICAL TRIAL: NCT01118221
Title: Rehabilitation of IPF Patients: Effects of Exercise and Oxidant Stress
Brief Title: Rehabilitation of Idiopathic Pulmonary Fibrosis (IPF) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O7467-R
Record Dates: First submitted 2010-04-27; First posted 2010-05-06 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: oxidant stress; exercise
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): enroll in pulmonary rehabilitation program
  Interventions: Behavioral: pulmonary rehabilitation
- Arm 2 (No Intervention): no structured exercise

INTERVENTIONS:
Behavioral: pulmonary rehabilitation — structured exercise program
  Arms: Arm 1

SUMMARY:
The incidence and prevalence of IPF increase exponentially with age, and IPF occurs more often in older males. Cigarette smoking and environmental dust exposures are known risk factors for developing IPF. For example, the recently deployed military population, as it ages, is at especially increased risk of IPF. No effective therapies exist, although lung transplantation is used to extend survival of selected patients.

Defining specific therapy to improve exercise tolerance and dyspnea in IPF patients is thus an urgent priority of veteran-oriented research programs.

DETAILED DESCRIPTION:
Chronic lung disease is common in the veteran population. While chronic obstructive pulmonary disease (COPD) is most prominent, fibrotic lung diseases, typified by idiopathic pulmonary fibrosis (IPF), are clearly increasing. We have developed extensive experience with a VA idiopathic pulmonary fibrosis (IPF) population in the context of a randomized, controlled clinical trial of vasodilator therapy.

Based on the current literature and our preliminary experience with exercise testing in IPF patients, we hypothesize that:

1. Formal pulmonary rehabilitation (i.e., an aerobic exercise program) will result in improved outcomes for IPF patients, demonstrable as an:

   1. Increase in exercise tolerance as quantified by 6-minute walk test (MWT) distance;
   2. Decrease in post-exercise dyspnea as quantified by the Borg dyspnea scale; and an
   3. Overall subjective improvement in quality of life as quantified by Saint George's Respiratory Questionnaire.
2. Metabolic and physiologic mechanisms of improved exercise tolerance and decreased dyspnea will include:

   1. More efficient oxygen metabolism demonstrated by maximum O2 uptake (VO2max);
   2. Decreased post-exercise oxidant stress demonstrated by post-exercise isoprostanes and plasma total antioxidant capacity (TAC); and,
   3. Maintenance of maximum inspiratory and expiratory pressures (PInmax and PExmax).

Our Specific Objectives are:

1. To investigate formal pulmonary rehabilitation and exercise tolerance in IPF patients

   The following important endpoints will be assessed to test the working hypothesis that pulmonary rehabilitation improves exercise capacity and lessens dyspnea:
   1. 6-MWT distance;
   2. Dyspnea index; and,
   3. Quality of life (Saint George's Respiratory Questionnaire [SGRQ] and International Physical Activity Questionnaire [IPAQ]).
2. To assess changes in oxygen uptake, markers of oxidant stress and pulmonary function resulting from pulmonary rehabilitation

To test the working hypothesis that improved outcomes are associated with more efficient O2 utilization, decreased markers of oxidant stress and maintained effort dependent pulmonary function, the following variables will be measured:

1. Peak oxygen uptake (VO2peak) during constant load exercise;
2. Markers of oxidant stress, including plasma and urine isoprostanes; and,
3. Maximum inspiratory and expiratory pressures (PInmax and PExmax). Completion of these Specific Objectives will position our research group to conduct future studies of 1) mechanisms of exercise limitation and 2) antioxidant therapies, both in this defined population and those who are at risk of developing pulmonary fibrosis. The long term impact of this application is thus to develop effective pulmonary rehabilitation strategies for IPF patients, based on knowledge of underlying changes in oxygen metabolism and oxidant stress.

ELIGIBILITY:
Inclusion Criteria:

* Clinical presentation consistent with IPF with onset between three months and 48 months prior to screening.
* Diagnosis made by high-resolution computed tomographic scan showing highly probable IPF.
* Absence of severe pulmonary hypertension (i.e., PAsys must be less than 55 mm Hg, based on echocardiography) and absence of decompensated right heart failure (NYHA class I or II acceptable).
* Age 40 through 80, inclusive.
* Abnormal pulmonary function tests (FVC 40-90% predicted or DLCO 30-90% predicted or impaired gas exchange with rest or exercise).
* Six-minute walk distance 150 m and 500 m.
* Worsening as demonstrated by any one of the following within the past year: > 10% decrease in percent predicted forced vital capacity or worsening dyspnea at rest or upon exertion, based on history.
* Ability to understand and sign a written informed consent form and comply with the requirements of the study.
* Absence of clinical features suggesting infection, neoplasm, sarcoidosis or collagen-vascular disease.

Exclusion Criteria:

* Echocardiographic evidence of severe pulmonary hypertension (PAsys>55 mm Hg, based on echocardiography or TR velocity 3.2 m/sec).
* Severe heart failure (NYHA class III or IV or LVEF < 45%).
* Six-minute walk distance < 150 m or > 500 m.
* FEV1/FVC ratio < 0.7 at screening (post-bronchodilator).
* Residual volume > 100% predicted.
* Any condition other than IPF likely to result in the death of the participant within the next two years.
* History of unstable or deteriorating cardiac or neurologic disease.
* Pregnancy or lactation. Patients who are: (a) pregnant or (b) breast feeding are excluded from the study.
* Current treatment with corticosteroids (either oral or inhaled), Cytoxan, azathioprine, colchicine, pirfenidone, anti-tumor necrosis factor therapy or endothelin receptor blockers. Prior treatment is permitted, but at least four weeks of treatment washout prior to inclusion in this study are required.
* Investigational therapy for any indication within 28 days prior to enrollment.
* Degenerative arthritis, cerebrovascular accident or other limitation to mobility preventing completion of the 6-minute walk test.
* Oxygen saturation on room air <80% at rest.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Jackson, MD, Principal Investigator — VA Medical Center, Miami
Locations (1):
- VA Medical Center, Miami, Miami, Florida, United States

REFERENCES:
- [Result] Jackson RM, Gomez-Marin OW, Ramos CF, Sol CM, Cohen MI, Gaunaurd IA, Cahalin LP, Cardenas DD. Exercise limitation in IPF patients: a randomized trial of pulmonary rehabilitation. Lung. 2014 Jun;192(3):367-76. doi: 10.1007/s00408-014-9566-9. Epub 2014 Apr 5. PMID 24705678
- [Result] Gaunaurd IA, Gomez-Marin OW, Ramos CF, Sol CM, Cohen MI, Cahalin LP, Cardenas DD, Jackson RM. Physical activity and quality of life improvements of patients with idiopathic pulmonary fibrosis completing a pulmonary rehabilitation program. Respir Care. 2014 Dec;59(12):1872-9. doi: 10.4187/respcare.03180. Epub 2014 Sep 2. PMID 25185149

RESULTS

PARTICIPANT FLOW:
Groups:
- Pulmonary Rehabilitation: enroll in pulmonary rehabilitation program
  pulmonary rehabilitation: structured exercise program
- Control: no structured exercise
Period: Overall Study
Arm/Group | Pulmonary Rehabilitation | Control
Started | 14 | 11
Completed | 11 | 10
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulmonary Rehabilitation | Control | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (6) | 66 (7) | 69 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 12 | 9 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 10 | 24
  South America | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: 6 Minute Walk Distance
Description: Change in 6 Minute Walk Distance from Baseline to 3 Months
Time Frame: The 6-MWD will be measured at 0 and 3 months.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 14 | 11
meters | -6.2 (86.9) | -15.3 (42.9)

2. Secondary Outcome: Systemic Markers of Oxidant Stress
Description: Plasma F2-isoprostanes measured in all subjects before and after exercise testing at baseline.
Time Frame: Markers of oxidant stress will be measured in all subjects before randomization after exercise testing at 0 months.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Before Exercise Testing: Plasma isoprostanes before exercise test.
- After Exercise Testing: Plasma isoprostanes after exercise testing.
Arm/Group | Before Exercise Testing | After Exercise Testing
Number analyzed (Participants) | 25 | 25
pg/mL | 16.48 (10.10) | 17.96 (10.05)

3. Secondary Outcome: Maximum Oxygen Uptake
Description: Change in 6 peak O2 uptake from Baseline to 3 Months
Time Frame: Maximum O2 uptake will be measured at 0 and 3 months.
Measure: Mean (Standard Error); unit: mL/minute
Groups:
- Rehabilitation Group: enroll in pulmonary rehabilitation program
  pulmonary rehabilitation: structured exercise program
- Control Group: no structured exercise
Arm/Group | Rehabilitation Group | Control Group
Number analyzed (Participants) | 14 | 11
mL/minute | -35 (71) | -119 (62)

ADVERSE EVENTS:
Time Frame: Six months.
Description: Adverse and unexpected events were recorded.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 0/14 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes